CLINICAL TRIAL: NCT01579097
Title: A Randomized, Comparative Phase 3 Trial to Assess the Safety and Efficacy of Triple-Chamber Parenteral Nutrition Formulation (Oliclinomel N4)
Brief Title: Comparative Phase 3 Trial to Assess the Safety and Efficacy of Triple-chamber Parenteral Nutrition Formulation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPIVTCHN001
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Nutrition Support
Keywords: (PN) Parenteral nutrition; oral/enteral not possible
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- compounded ternary parenteral nutrition (Active Comparator): compounded ternary Parenteral Nutrition admixture
  Interventions: Other: Compounded ternary parenteral nutrition admixtures
- Oliclinomel N4 formulation (Experimental): Oliclinomel N4 is a ready-to-use PN product presented as a triple chamber bag
  Interventions: Other: Oliclinomel N4

INTERVENTIONS:
Other: Oliclinomel N4 — Oliclinomel is a PN product which provides the macronutrients (e.g., dextrose, amino acids, and lipids) for patients when oral or enteral nutrition is not possible, insufficient, or contraindicated
  Other Names: Oliclinomel N4-550
  Arms: Oliclinomel N4 formulation
Other: Compounded ternary parenteral nutrition admixtures — Study treatment will be administered for a minimum of 5 days up to a maximum of 14 days
  Arms: compounded ternary parenteral nutrition

SUMMARY:
The objective of this study is to assess the safety and efficacy of Oliclinomel N4 compared to compounded ternary parenteral nutrition (PN) admixtures for the delivery of PN in hospitalized adults for whom oral or enteral nutrition is not possible, insufficient, or contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient but hospitalized < 14 days prior to enrollment
* Requires PN because oral or enteral nutrition is not possible, insufficient, or contraindicated
* Has capability to complete at least 5 days of study treatment (i.e., PN)
* Has a useable peripheral vein for delivery of intravenous (IV) PN

Exclusion Criteria:

* Has a life expectancy of < 6 days from initiation of study treatment, in the opinion of the Investigator
* Known hypersensitivity to the components of either of the investigational study treatments
* Use of prohibited medications (e.g. glucocorticosteroids or antitumor chemotherapeutic agents) within 30 days prior to enrollment
* Known serious clinically significant condition that would preclude participation in the study
* Known chronic active hepatitis, elevated liver function tests
* Known history of human immunodeficiency virus infection
* Known severe dyslipidemia, severe hyperglycemia,clinically significant abnormalities of plasma electrolytes
* Known pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Serum Prealbumin | Serum Prealbumin at Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Baxter Investigative Site, Study Director — Shanghai, China; Baxter Investigative Site, Study Director — Shantou, China; Baxter Investigative Site, Study Director — Haikou, China; Baxter Investigative Site, Study Director — Jiangsu Province, China; Baxter Investigative Site, Study Director — Beijing, China; Baxter Investigative Site, Study Director — Changsha, China; Baxter Investigative Site, Study Director — Hangzhou, China; Baxter Investigative Site, Study Director — Nanning, China; Baxter Investigative Site, Study Director — Shang dong Province, China
Locations (1):
- Shanghai No. 6 Hospital, Shanghai, China